CLINICAL TRIAL: NCT01433328
Title: Lidocaine Subcutaneous Infusion for Control of Treprostinil Related Site Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Safety considerations
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr David Langleben, Chair, Cardiology Department, Jewish General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JGH-11-096
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Remodulin; Treprostinil
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental)
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Remodulin only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Lidocaine
  Arms: Lidocaine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Treprostinil subcutaneous (under the skin) infusion is a very good medication for treating pulmonary arterial hypertension but infusion site pain may be very severe in some patients. The investigators plan to treat patients receiving treprostinil with a subcutaneous infusion of lidocaine (a local anesthestic) to treat the pain.

ELIGIBILITY:
Inclusion Criteria:

* PAH
* Treprostinil treatment for at least 3 months
* Severe infusion site pain

Exclusion Criteria:

* Pregnancy/breastfeeding
* Decompensated heart failure
* Chronic liver disease
* Abnormal electrolytes
* Heart block (2/3 degree), sino-atrial block, idioventricular rhythm
* Systolic systemic BP <90mmHg
* Bradycardia HR <55
* Adverse reaction to lidocaine or other amide local anesthestic
* Interacting medications (anti-arrhythmics, CYP1A2 inhibitors)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pain Questionnaire | 1 week
  Short Form McGill Pain Questionnaire - Change from baseline over one week
Daily Pain Diary | 1 week
  10cm visual analogue scale (VAS) - Change in aggregated median/maximum scores over one week

SECONDARY OUTCOMES:
proNT-BNP | 1 week
6 minute walk | 1 week
Lidocaine level | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: David Langleben, MD, Principal Investigator — Chair, Cardiology Department
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada